CLINICAL TRIAL: NCT02827045
Title: Exploratory Study of a Vestibular Biomarker of Phase in Bipolar Disorder
Brief Title: Study of a Vestibular Biomarker of Phase in Bipolar Disorder
Acronym: BDmarker
Status: Enrolling by invitation | Type: Observational
Sponsor: Vest Brain,Centro de Estudios Neurovestibulares (Other)
Responsible Party: Principal Investigator, Ana Maria Soza Ried, Dr., Vest Brain,Centro de Estudios Neurovestibulares
Other Study IDs: VESTBRAIN002
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Bipolar Disorder; Depression, Bipolar
MeSH Terms: conditions — Bipolar Disorder | interventions — Vestibular Function Tests

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Depressive phase: Vestibular test
  Interventions: Device: Vestibular test
- Maniac phase: Vestibular test
  Interventions: Device: Vestibular test
- Euthimic phase: Vestibular test
  Interventions: Device: Vestibular test
- Healthy subject: Vestibular test
  Interventions: Device: Vestibular test

INTERVENTIONS:
Device: Vestibular test

SUMMARY:
Bipolar Disorder show cyclic changes of mood between depression (depressive phase) and mania (maniac phase). Vestibular tests have been shown high sensibility and specificity as a biological marker for major depression. This exploratory investigation will measure and compare the vestibular activity of bipolar disorder patients during different phases ( 6 depressed phase, 6 maniac phase, 6 euthimic and 6 control healthy subjects).

ELIGIBILITY:
Inclusion Criteria:

* Bipolar disorder I or II
* depressive phase of bipolar disorder
* maniac phase of bipolar disorder
* euthimic phase of bipolar disorder

Exclusion Criteria:

* drugs addiction
* alcohol addiction
* neurologic condition, disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: study population come from psychiatric care consults
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2016-07; Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Vestibular test | December 2017

IPD SHARING:
Plan to Share IPD: No